CLINICAL TRIAL: NCT02730377
Title: Efficacy in Controlling Glycaemia With Victoza® (Liraglutide) as add-on to Metformin vs. OADs as add-on to Metformin After up to 104 Weeks of Treatment in Subjects With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy and Treated in a Primary Care Setting
Brief Title: Efficacy in Controlling Glycaemia With Victoza® (Liraglutide) as add-on to Metformin vs. OADs as add-on to Metformin After up to 104 Weeks of Treatment in Subjects With Type 2 Diabetes
Acronym: LIRA-PRIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-4232; 2015-002417-29 (EudraCT Number); U1111-1170-7035 (Other: WHO)
Record Dates: First submitted 2016-03-23; First posted 2016-04-06 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Glycoside Hydrolase Inhibitors; Dipeptidyl-Peptidase IV Inhibitors; meglitinide; Sodium-Glucose Transporter 2 Inhibitors; Sulfonylurea Compounds; Thiazolidinediones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide 1.8 mg (Experimental): Add-on to metformin
  Interventions: Drug: liraglutide
- OAD (Active Comparator): Add-on to metformin. Treatment with one OAD selected at the discretion of the investigator. Subjects randomised to the OAD arm must remain on the same OAD throughout the trial.
  Interventions: Drug: alpha-glucosidase inhibitors; Drug: DPP-4 inhibitors; Drug: meglitinides; Drug: SGLT-2 inhibitors; Drug: sulphonylurea; Drug: thiazolidinediones

INTERVENTIONS:
Drug: liraglutide — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: Liraglutide 1.8 mg
Drug: alpha-glucosidase inhibitors — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD
Drug: DPP-4 inhibitors — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD
Drug: meglitinides — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD
Drug: SGLT-2 inhibitors — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD
Drug: sulphonylurea — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD
Drug: thiazolidinediones — Trial product will be prescribed by the investigator and dispensed by pharmacy or similar.
  Arms: OAD

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate efficacy in controlling glycaemia with Victoza® (liraglutide) as add-on to metformin background treatment vs. OADs as add-on to metformin background treatment for 104 weeks of treatment in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Male or female at least 18 years of age at the time of signing informed consent - Subjects diagnosed (clinically) with type 2 diabetes equal to or above 90 days prior to the screening visit - Stable daily dose of metformin as monotherapy equal to or above 1500 mg or maximum tolerated dose within 60 days prior to the screening visit - HbA1c 7.5-9.0% (59-75 mmol/mol) (both inclusive) and measured within the last 90 days prior to the screening visit Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) - Treatment with any medication for the indication of diabetes other than metformin in a period of 60 days before the screening visit. An exception is short-term treatment (below or equal to 7 days in total) with insulin in connection with intercurrent illness - Receipt of any investigational medicinal product within 30 days before the screening visit - Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1991 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (201):
- United States (160):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Haleyville, Alabama
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Fountain Hills, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Harrisburg, Arkansas
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, North Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Alhambra, California
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Carlsbad, California
  - Novo Nordisk Investigational Site, Coronado, California
  - Novo Nordisk Investigational Site, Costa Mesa, California
  - Novo Nordisk Investigational Site, Elk Grove, California
  - Novo Nordisk Investigational Site, Encinitas, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Mirada, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Oxnard, California
  - Novo Nordisk Investigational Site, Rancho Cucamonga, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Westminster, California
  - Novo Nordisk Investigational Site, Centennial, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Monument, Colorado
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Ocoee, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Ormond Beach, Florida
  - Novo Nordisk Investigational Site, Oviedo, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Seminole, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Bainbridge, Georgia
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Perry, Georgia
  - Novo Nordisk Investigational Site, Statesboro, Georgia
  - Novo Nordisk Investigational Site, Suwanee, Georgia
  - Novo Nordisk Investigational Site, Woodstock, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Aurora, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gillespie, Illinois
  - Novo Nordisk Investigational Site, Wauconda, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Newton, Kansas
  - Novo Nordisk Investigational Site, Park City, Kansas
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Sunset, Louisiana
  - Novo Nordisk Investigational Site, Elkridge, Maryland
  - Novo Nordisk Investigational Site, Oxon Hill, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Rochester, Michigan
  - Novo Nordisk Investigational Site, Sterling Heights, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Belzoni, Mississippi
  - Novo Nordisk Investigational Site, Port Gibson, Mississippi
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Missoula, Montana
  - Novo Nordisk Investigational Site, Fremont, Nebraska
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, Westfield, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Burlington, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Elizabeth City, North Carolina
  - Novo Nordisk Investigational Site, Garner, North Carolina
  - Novo Nordisk Investigational Site, Mooresville, North Carolina
  - Novo Nordisk Investigational Site, Morganton, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Edmond, Oklahoma
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Fleetwood, Pennsylvania
  - Novo Nordisk Investigational Site, Harleysville, Pennsylvania
  - Novo Nordisk Investigational Site, Jersey Shore, Pennsylvania
  - Novo Nordisk Investigational Site, Lansdale, Pennsylvania
  - Novo Nordisk Investigational Site, Levittown, Pennsylvania
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Smithfield, Pennsylvania
  - Novo Nordisk Investigational Site, Uniontown, Pennsylvania
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Old Point Station, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Athens, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Humboldt, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Tullahoma, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Georgetown, Texas
  - Novo Nordisk Investigational Site, Gonzales, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Kerrville, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Missouri City, Texas
  - Novo Nordisk Investigational Site, New Braunfels, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Splendora, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Bountiful, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Danville, Virginia
  - Novo Nordisk Investigational Site, Gloucester Courthouse, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Bellevue, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Walla Walla, Washington
- Canada (11):
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Truro, Nova Scotia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Strathroy, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - Novo Nordisk Investigational Site, Québec
- Colombia (2):
  - Novo Nordisk Investigational Site, Bogotá
  - Novo Nordisk Investigational Site, Medellín
- India (11):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Nagpur, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Hyderabad, Telangana
  - Novo Nordisk Investigational Site, Lucknow, Uttar Pradesh
  - Novo Nordisk Investigational Site, Noida, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hubli
  - Novo Nordisk Investigational Site, Ludhiana
- Latvia (2):
  - Novo Nordisk Investigational Site, Riga
  - Novo Nordisk Investigational Site, Tukums
- Lebanon (4):
  - Novo Nordisk Investigational Site, Beirut
  - Novo Nordisk Investigational Site, Byblos
  - Novo Nordisk Investigational Site, El Achrafiyé
  - Novo Nordisk Investigational Site, Hazmiyeh
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Toa Baja
  - Novo Nordisk Investigational Site, Trujillo Alto
- Russia (3):
  - Novo Nordisk Investigational Site, Dzerzhinskiy
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Serbia (4):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Adapazarı
  - Novo Nordisk Investigational Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Background] Unger J, Allison DC, Carlton M, Lakkole K, Lowe D, Murphy G, Panda JK, Sargin M, Kaltoft M, Treppendahl MB, Zoghbi M; LIRA-PRIME global panel. Trial design and baseline data for LIRA-PRIME: A randomized trial investigating the efficacy of liraglutide in controlling glycaemia in type 2 diabetes in a primary care setting. Diabetes Obes Metab. 2019 Jul;21(7):1543-1550. doi: 10.1111/dom.13682. Epub 2019 Mar 26. PMID 30828917
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 219 sites in Canada (11), Colombia (3), India (16), Latvia (2), Lebanon (4), Russian Federation (5), Serbia (6), Turkey (4) and the United States (168).
Pre-assignment Details: Participants were randomised in a 1:1 manner to receive either liraglutide or an oral antidiabetic drug (OAD) both as add-on to background therapy with metformin.
Groups:
- Liraglutide 1.8 mg: Participants were to receive a subcutaneous injection of liraglutide once daily. Participants received 0.6 milligrams (mg) liraglutide during the first week. The dose was escalated in weekly increments of 0.6 mg until the dose of 1.8 mg was reached. The treatment period was 104 weeks.
- Oral Antidiabetic Drug: Participants were to receive one selected OAD. The following OADs were allowed: alpha-glucosidase inhibitors, dipeptidyl peptidase-4 (DPP-4) inhibitors, meglitinides, sodium-glucose co-transporter-2 (SGLT-2) inhibitors, sulfonylureas or thiazolidinediones. The treatment period was 104 weeks.
Period: Overall Study
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Started | 996 | 995
Treated | 980 | 984
Full Analysis Set (FAS) | 996 | 995
Safety Analysis Set (SAS) | 980 | 984
Completed | 446 | 362
Not Completed | 550 | 633
Not completed — Other | 5 | 4
Not completed — Death | 1 | 8
Not completed — Inadequate glycaemic control | 368 | 473
Not completed — Adverse Event | 79 | 41
Not completed — Protocol Violation | 23 | 30
Not completed — Lack of Efficacy | 4 | 13
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 45 | 42
Not completed — Lost to Follow-up | 25 | 21

BASELINE CHARACTERISTICS:
Population: FAS included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug | Total
Number analyzed (Participants) | 996 | 995 | 1991
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (11.0) | 57.1 (10.7) | 57.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 476 | 471 | 947
  Male | 520 | 524 | 1044
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 176 | 189 | 365
  Not Hispanic or Latino | 820 | 806 | 1626
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 3 | 6 | 9
    Asian | 149 | 141 | 290
    Black or African American | 101 | 106 | 207
    Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
    White | 724 | 714 | 1438
    Other | 16 | 26 | 42

OUTCOME MEASURES:

1. Primary Outcome: Time to Inadequate Glycaemic Control
Description: Inadequate glycaemic control was defined as glycosylated haemoglobin (HbA1c) of 7.0% (53 mmol/mol) or greater at two consecutive visits after the first 26 weeks of treatment and up to 104 weeks. 25%, median (50%) and 75% percentiles for the cumulative distribution function, are obtained from the Kaplan-Meier survival function. HbA1c was recorded at weeks 38, 52, 65, 78, 91 and 104.
Time Frame: Weeks 26-104
Population: FAS included all randomised participants. Overall number of participants analyzed=participants with available data.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 416 | 547
Weeks | 108.9 [37.7 to NA] — The 75 percentile data was not available as the proportion was not reached within study period. | 64.9 [35.4 to 107.4]
Statistical Analysis 1: Comparison: Liraglutide 1.8 mg vs Oral Antidiabetic Drug; Test for no treatment difference is based on using a generalised log-rank test for interval censored failure time data; Test type: Superiority; p < .0001, Log Rank

2. Secondary Outcome: Time to Premature Treatment Discontinuation (for Any Reason Including Inadequate Glycaemic Control)
Description: The time to premature treatment discontinuation (for any reason including inadequate glycaemic control) was analysed and presented using the generalised log rank test. 25%, median (50%) and 75% percentiles for the cumulative distribution function, are obtained from the Kaplan-Meier survival function.
Time Frame: Weeks 0-104
Population: FAS included all randomised participants. Overall number of participants analyzed=participants with available data.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 532 | 624
Weeks | 80.4 [35.7 to NA] — The 75 percentile data was not available as the proportion was not reached within study period. | 52.3 [35.1 to NA] — The 75 percentile data was not available as the proportion was not reached within study period.

3. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in HbA1c at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: Overall number of participants analyzed=FAS included all randomised participants. Number analyzed=participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Percentage point of HbA1c
  Change at week 104: number analyzed (Participants) | 404 | 327
  Change at week 104 | -1.4 (1.06) | -1.1 (1.04)
  Change at premature treatment discontinuation: number analyzed (Participants) | 108 | 79
  Change at premature treatment discontinuation | -0.6 (1.03) | -0.2 (1.56)

4. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (Yes/No)
Description: Participants who achieved HbA1c ≤6.5% (yes/no) is presented.
Time Frame: Week 104/Premature treatment discontinuation
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Participants
  Yes | 255 | 162
  No | 741 | 833

5. Secondary Outcome: Participants Who Achieve HbA1c ≤7.0% Without Weight Gain
Description: Participants who achieved HbA1c ≤7.0% without weight gain (yes/no) is presented.
Time Frame: Week 104/Premature treatment discontinuation
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Participants
  Yes | 329 | 234
  No | 667 | 761

6. Secondary Outcome: Participants Who Achieve HbA1c ≤7.0% Without Treatment Emergent Severe Hypoglycaemic Episodes or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value <3.1 millimoles per liter (mmol/L) with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than the day after the last day on trial product. Participants who achieved HbA1c ≤7.0% without treatment emergent severe hypoglycaemic episodes or BG confirmed symptomatic hypoglycaemic episodes (yes/no) is presented.
Time Frame: Week 104/Premature treatment discontinuation
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Participants
  Yes | 388 | 292
  No | 608 | 703

7. Secondary Outcome: Participants Who Achieve HbA1c ≤7.0% Without Weight Gain and no Treatment Emergent Severe Hypoglycaemic Episodes or Blood Glucose Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than the day after the last day on trial product. Participants who achieved HbA1c ≤7.0% without weight gain and no treatment emergent severe hypoglycaemic episodes or BG confirmed symptomatic hypoglycaemic episodes (yes/no) is presented.
Time Frame: Week 104/Premature treatment discontinuation
Population: FAS included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Participants
  Yes | 320 | 227
  No | 676 | 768

8. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Millimoles per liter (mmol/L)
  Change at week 104: number analyzed (Participants) | 418 | 346
  Change at week 104 | -2.2 (2.65) | -1.2 (2.46)
  Change at premature treatment discontinuation: number analyzed (Participants) | 103 | 78
  Change at premature treatment discontinuation | -0.6 (2.91) | -0.6 (3.76)

9. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Kilogram (Kg)
  Change at week 104: number analyzed (Participants) | 427 | 349
  Change at week 104 | -3.8 (6.38) | -3.5 (6.19)
  Change at premature treatment discontinuation: number analyzed (Participants) | 116 | 86
  Change at premature treatment discontinuation | -2.9 (3.74) | -2.2 (4.93)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) in BMI at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Kilograms per square meter (kg/m^2)
  Change at week 104: number analyzed (Participants) | 427 | 349
  Change at week 104 | -1.3 (2.26) | -1.2 (2.14)
  Change at premature treatment discontinuation: number analyzed (Participants) | 116 | 86
  Change at premature treatment discontinuation | -1.1 (1.33) | -0.8 (1.71)

11. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change from baseline (week 0) in systolic and diastolic blood pressure at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 996 | 995
Millimeters of mercury (mmHg)
  SBP: Change at week 104: number analyzed (Participants) | 429 | 350
  SBP: Change at week 104 | -2.4 (15.09) | -1.1 (15.11)
  SBP: Change at premature treatment discontinuation: number analyzed (Participants) | 117 | 87
  SBP: Change at premature treatment discontinuation | -2.8 (15.99) | -2.9 (15.23)
  DBP: Change at week 104: number analyzed (Participants) | 429 | 351
  DBP: Change at week 104 | -1.3 (9.51) | -0.6 (9.54)
  DBP: Change at premature treatment discontinuation: number analyzed (Participants) | 117 | 87
  DBP: Change at premature treatment discontinuation | -1.0 (11.27) | 0.2 (9.69)

12. Secondary Outcome: Number of Severe Hypoglycaemic Episodes
Description: Severe hypoglycaemic episodes were defined as episodes that required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Number of severe hypoglycaemic episodes that occured during weeks 0-104 are presented.
Time Frame: Weeks 0-104
Population: Safety analysis set (SAS) included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Episodes | 32 | 52

13. Secondary Outcome: Number of Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Number of severe or BG confirmed symptomatic hypoglycaemic episodes that occured during weeks 0-104 are presented.
Time Frame: Weeks 0-104
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Episodes | 24 | 44

14. Secondary Outcome: Number of Documented Symptomatic Hypoglycaemic Episodes (ADA)
Description: Documented symptomatic hypoglycaemic were defined as episodes with typical symptoms of hypoglycaemia accompanied by measure plasma glucose concentration <= 3.9 mmol/L. Number of documented symptomatic hypoglycaemic episodes that occured during the weeks 0-104 are presented.
Time Frame: Weeks 0-104
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Episodes | 98 | 155

15. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was defined as any event that resulted in any of the following: death, life-threatening experience, in-patient hospitalisation or prolongation of existing hospitalisation, persistent or significant disability or incapacity, congenital anomaly or birth defect or suspicion of transmission of infectious agents via the trial product. An SAE was considered as treatment emergent if it had an onset or increase in severity on or after the time of first trial product administration and no later than 7 days after the time of last trial product administration. Number of treatment emergent serious adverse events are presented.
Time Frame: Weeks 0-105
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Events | 145 | 140

16. Secondary Outcome: Number of AEs Leading to Permanent Discontinuation of Trial Product
Description: An adverse event (AE) was any untoward medical occurrence in a participant who administered a product, and which did not necessarily had a causal relationship with this treatment. An AE was considered as treatment emergent if it had an onset or increase in severity on or after the time of first trial product administration and no later than 7 days after the time of last trial product administration. Number of treatment emergent AEs that led to permanent discontinuation of trial product are presented.
Time Frame: Weeks 0-105
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Events | 188 | 98

17. Secondary Outcome: Change in Lipids: HDL Cholesterol, LDL-cholesterol, Total Cholesterol, Triglycerides
Description: Change from baseline (week 0) in high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, total cholesterol (TC) and triglycerides (TG) at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: Overall number of participants analyzed=SAS included all participants exposed to at least one dose of trial product. Number analyzed=participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Millimoles per liter (mmol/L)
  HDL: Change at week 104: number analyzed (Participants) | 417 | 339
  HDL: Change at week 104 | 0.1 (0.20) | 0.1 (0.19)
  HDL: Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  HDL: Change at premature treatment discontinuation | -0.0 (0.17) | 0.0 (0.20)
  LDL: Change at week 104: number analyzed (Participants) | 417 | 339
  LDL: Change at week 104 | -0.1 (0.80) | 0.0 (0.83)
  LDL: Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  LDL: Change at premature treatment discontinuation | -0.1 (0.68) | -0.1 (0.85)
  TC: Change at week 104: number analyzed (Participants) | 419 | 340
  TC: Change at week 104 | -0.2 (0.92) | 0.1 (0.99)
  TC: Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  TC: Change at premature treatment discontinuation | -0.0 (0.81) | -0.1 (0.96)
  TG: Change at week 104: number analyzed (Participants) | 418 | 340
  TG: Change at week 104 | -0.3 (0.95) | -0.1 (1.25)
  TG: Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  TG: Change at premature treatment discontinuation | -0.0 (1.13) | -0.0 (1.30)

18. Secondary Outcome: Change in Biochemistry- Alanine Aminotransferase (ALAT), Amylase, Aspartate Aminotransferase (ASAT), Lipase
Description: Change from baseline (week 0) in alanine aminotransferase (ALAT), amylase, aspartate aminotransferase (ASAT) and lipase at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Units per liter (U/L)
  ALAT: Week 104: number analyzed (Participants) | 408 | 331
  ALAT: Week 104 | -4.6 (17.83) | -5.4 (17.13)
  ALAT: Premature treatment discontinuation: number analyzed (Participants) | 107 | 79
  ALAT: Premature treatment discontinuation | -3.2 (12.44) | -3.3 (14.67)
  Amylase: Week 104: number analyzed (Participants) | 419 | 340
  Amylase: Week 104 | 8.9 (30.93) | 5.1 (26.30)
  Amylase: Premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  Amylase: Premature treatment discontinuation | 0.6 (23.61) | 2.1 (17.92)
  ASAT: Week 104: number analyzed (Participants) | 409 | 337
  ASAT: Week 104 | -2.0 (13.27) | -2.3 (11.85)
  ASAT: Premature treatment discontinuation: number analyzed (Participants) | 108 | 79
  ASAT: Premature treatment discontinuation | -1.9 (10.76) | -0.4 (11.64)
  Lipase: Week 104: number analyzed (Participants) | 419 | 340
  Lipase: Week 104 | 15.1 (67.69) | -0.5 (50.03)
  Lipase: Premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  Lipase: Premature treatment discontinuation | 10.4 (32.40) | -2.2 (35.79)

19. Secondary Outcome: Change in Biochemistry- Creatinine, Total Bilirubin
Description: Change from baseline (week 0) in creatinine and total bilirubin (TB) at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Micromoles per liter (umol/L)
  Creatinine: week 104: number analyzed (Participants) | 419 | 340
  Creatinine: week 104 | 3.3 (13.37) | 1.0 (12.86)
  Creatinine: premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  Creatinine: premature treatment discontinuation | 2.9 (12.06) | 2.6 (21.13)
  TB: week 104: number analyzed (Participants) | 408 | 331
  TB: week 104 | 0.4 (4.47) | 0.7 (3.80)
  TB: premature treatment discontinuation: number analyzed (Participants) | 107 | 79
  TB: premature treatment discontinuation | -0.0 (2.78) | -0.6 (3.17)

20. Secondary Outcome: Change in Biochemistry- Estimated Glomerular Filtration Rate (eGFR) Serum
Description: The estimated GFR was derived from serum creatinine using the MDRD (Modification of diet in renal disease) formula. eGFR was measured as milliliter per min per specific surface area (mL/min/SSA).
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mL/min/SSA
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
mL/min/SSA
  Change at week 104: number analyzed (Participants) | 419 | 340
  Change at week 104 | -5.1 (20.33) | -1.6 (16.29)
  Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  Change at premature treatment discontinuation | -3.0 (12.56) | -1.7 (15.01)

21. Secondary Outcome: Change in Potassium
Description: Change from baseline (week 0) in potassium at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Millimoles per liter (mmol/L)
  Change at week 104: number analyzed (Participants) | 419 | 339
  Change at week 104 | -0.1 (0.60) | -0.0 (0.59)
  Change at premature treatment discontinuation: number analyzed (Participants) | 109 | 80
  Change at premature treatment discontinuation | -0.0 (0.44) | -0.2 (0.71)

22. Secondary Outcome: Change in Haemoglobin
Description: Change from baseline (week 0) in haemoglobin at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Grams per deciliter (g/dL)
  Change at week 104: number analyzed (Participants) | 399 | 331
  Change at week 104 | -0.4 (1.07) | -0.0 (1.16)
  Change at premature treatment discontinuation: number analyzed (Participants) | 105 | 76
  Change at premature treatment discontinuation | -0.3 (0.87) | -0.3 (1.12)

23. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) in pulse at week 104 or at premature treatment discontinuation is presented.
Time Frame: Week 0, week 104/premature treatment discontinuation
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
Number analyzed (Participants) | 980 | 984
Beats per minute (beats/min)
  Change at week 104: number analyzed (Participants) | 429 | 350
  Change at week 104 | 1.0 (10.25) | -0.6 (10.23)
  Change at premature treatment discontinuation: number analyzed (Participants) | 115 | 86
  Change at premature treatment discontinuation | 0.7 (9.84) | 0.9 (10.59)

ADVERSE EVENTS:
Time Frame: Weeks 0-105
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product administration. Results are based on the SAS which included all participants exposed to at least one dose of trial product.
Arm/Group | Liraglutide 1.8 mg | Oral Antidiabetic Drug
All-Cause Mortality (participants affected / at risk) | 1/980 | 8/984
Serious Adverse Events (participants affected / at risk) | 92/980 | 81/984
Other Adverse Events (participants affected / at risk) | 65/980 | 15/984
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=980) | Oral Antidiabetic Drug (N=984)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (7) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 6 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 4 (4) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 4 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Empty sella syndrome (Endocrine disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Exophthalmos (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 2 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 1.8 mg (N=980) | Oral Antidiabetic Drug (N=984)
Nausea (Gastrointestinal disorders) | 65 (82) | 15 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02730377/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02730377/SAP_001.pdf